CLINICAL TRIAL: NCT01674114
Title: Postoperative Morphine Consumption After Caesarean Section- TAP Block vs Intracutaneous Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-1
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy
Keywords: Cesarean Section; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (Experimental): transversus abdominis plane block (TAP block). Ultrasound guided TAP-block at the end of surgery using 20 ml bupivacaine 0,25% with Adrenaline 5mcg/ml bilaterally by the anaesthesiologist, and 20 ml NaCl intracutaneously in the operating wound performed by the obstetrician
  Interventions: Procedure: TAP block
- control (Active Comparator): Ultrasound guided TAP block at the end of surgery with 20 ml NaCl bilaterally and 20 ml bupivacaine 0,25% with Adrenaline 5mcg/ml intracutaneously in the surgical wound(standard practice)
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: TAP block
  Arms: TAP block
Procedure: control
  Other Names: intracutaneous infiltration
  Arms: control

SUMMARY:
The purpose of this study is to investigate whether a regional-block (TAP block) in Caesarean section will give a measurable benefit in form of reducing Morphine consumption as compared to local infiltration of the wound with local anesthetic.

DETAILED DESCRIPTION:
Caesarean section is one of the most common surgical procedures in the world and postoperative pain afflicts both mother and the newborn- especially the first 48 hours after birth.

Pain management at the investigators hospital is multimodal (balanced analgesia). Peroperatively the wound is infiltrated with local anaesthetic performed by the obstetrician at the end of the procedure. Postoperatively the patient gets routinely a combination of Paracetamol and NSAID's orally and Morphine intravenously as required. The side-effects of Morphine (nausea, vomiting, itching and sedation) do interfere, dose dependent, with the interaction between mother and child, breastfeeding and postpartum experience.

Previous studies have compared transversus abdominis plane block (TAP block) with reduction of morphine consumption in C-section (up to 50%! (1,2). So far no one has compared TAP-block with local infiltration in C-section patients.

Ultrasound guided TAP-block is done by an anaesthesiologist at the end of the operation, and it is viewed as a safe and easy procedure to perform. The investigators assumption is that the TAP-block reduces the morphine consumption with 50% as compared to local infiltration. Due to maximal dosage of Bupivacaine, it is not possible to give both types of anaesthesia at the same time.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women that are scheduled for elective C-section

Exclusion Criteria:

* relevant drug allergy
* history of drug abuse

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
total amount of morphine consumption | 48 hours
  patient controlled analgesia (PCA-pump)

SECONDARY OUTCOMES:
time to first bolus request | up to 48 hours
cumulative morphine consumption | 12 hours
cumulative morphine consumption | 24 hours
cumulative morphine consumption | 36 hours
pain | up to 48 hours
  Visual Analog Scale 0-10
side effects | up to 48 hours
  nausea, vomiting, pruritus and sedation on a 4 point scale as none, mild, moderate and severe

OTHER OUTCOMES:
anti-emetics | up to 48 hours
  Antiemetics will not be given routinely, and its use will therefore also be registered

CONTACTS AND LOCATIONS:
Overall Officials: Aage Telnes, MD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Telnes A, Skogvoll E, Lonnee H. Transversus abdominis plane block vs. wound infiltration in Caesarean section: a randomised controlled trial. Acta Anaesthesiol Scand. 2015 Apr;59(4):496-504. doi: 10.1111/aas.12498. PMID 25786679